CLINICAL TRIAL: NCT04460833
Title: Feedback in Augmented Reality to Control the Gait Parameters in Children With Cerebral Palsy (BestOf_ARRoW)
Brief Title: Feedback in Augmented Reality to Control of Gait Parameters in Children With Cerebral Palsy
Acronym: BestOf_ARRoW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ellen Poidatz (Other)
Collaborators: Université Paris-Sud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BestOf_ARRoW Feedback
Record Dates: First submitted 2020-03-12; First posted 2020-07-08 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy; Gait Disorders, Neurologic; Feedback, Psychological
Keywords: Serious Game; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Masking Description: Feedback modalities are given through an augmented reality headset by random
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): All children will have the 6 feedback modalities + the control given randomly
  Interventions: Device: Feedback modalities given through an augmented reality headset

INTERVENTIONS:
Device: Feedback modalities given through an augmented reality headset — All children wear the augmented reality headset. After a habituation period to the holograms, they start the protocol. It consists of a warm-up session, training session (which three feedback modalities are presented), calibration session (to get the maximal speed and spontaneous speed of the child), and test session. During test session, all the children walk on the 30m corridor. They have 6 feedback modalities + the control, given randomly. On the way out, they have to walk fast as possible ; on the return they have to walk at intermediate speed.

SUMMARY:
Cerebral palsy (CP) describes a group of permanent disorders of the development of movement and posture, causing activity limitation, that are attributed to non progressive disturbances that occurred in the developing fetal or infant brain. The motor disorder of CP are often accompanied by disturbances of sensation, perception, cognition, communication, and behaviour; by epilepsy, and by secondary musculoskeletal problems.

Motor activities, especially walking, can be affected by many factors including sensory deficits, biomechanical and postural limitations, muscle weakness and spasticity.To provide feedback, during gait rehabilitation is a complementary approach to improve motor learning during the rehabilitation protocol. However, the feedback modalities are multiple and no study has compared these modalities. This study aims to test which feedback modalities could control the gait parameters (speed, cadence, step length) of the child with CP in real-time, through an augmented reality environment.

ELIGIBILITY:
Inclusion Criteria:

* Children with Cerebral palsy (medical file)
* Age 12-18
* Global Motor Function Classification System (GMFCS) I-III
* Functional Mobility Scale (FMS) minimum 2 for "50 meters"
* Ability to cooperate, to understand and to follow instructions
* Patient affiliated to the French social security system
* Patient volunteers whose the parents given their authorization to participate

Exclusion Criteria:

* Medical decision for any reason
* Child or parent decision for any reason
* Inability to cooperate, to understand and to follow instructions

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
walking speed | 1 year
  Walking speed recorded with the augmented reality headset in real-time
step length | 1 year
  step length recorded with the augmented reality headset in real-time

SECONDARY OUTCOMES:
Moizer Questionary | 1 year
  User experience survey; 25 items scored 1 for "I perfectly agree" to 5 "I completly disagree" this item; max score = 25; min score = 125

CONTACTS AND LOCATIONS:
Overall Officials: Eric DESAILLY, PhD, Principal Investigator — Fondation Ellen Poidatz
Locations (1):
- Fondation Ellen Poidatz, Saint-Fargeau-Ponthierry, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guinet AL, Bouyer G, Otmane S, Desailly E. Visual Feedback in Augmented Reality to Walk at Predefined Speed Cross-Sectional Study Including Children With Cerebral Palsy. IEEE Trans Neural Syst Rehabil Eng. 2022;30:2322-2331. doi: 10.1109/TNSRE.2022.3198243. Epub 2022 Aug 22. PMID 35951576
- See also: Website of the EllenPoidatz Foundation (See Research and Innovation) — https://www.fondationpoidatz.com/